CLINICAL TRIAL: NCT06150053
Title: Dose Dense Chemotherapy in Elderly Patients > 80 Years Old With DLBCL
Status: Completed | Type: Observational
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Konstantinos Christofyllakis, Consultant, University Hospital, Saarland
Organization: Universität des Saarlandes (Other)
Other Study IDs: DOME-80
Record Dates: First submitted 2022-05-05; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: DLBCL; Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- R-CHOP-14
- R-mini-CHOP

SUMMARY:
Multi-center retrospective analysis of patients with DLBCL aged ≥80 years old treated with R-CHOP-14 compared to other regimens. Patient data including baseline characteristics, histology, dose intensity and treatment outcomes will be extracted from hospital medical electronic records. Relative dose intensity (RDI) will be calculated as the percentage of the dose intensity achieved divided by the intended dose intensity. Primary endpoints are overall (OS), progression-free (PFS) and event-free survival (EFS), defined as time from diagnosis to death, death or progression/relapse, progression/relapse or treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven, untreated diffus large B-cell lymphoma (DLBCL)
* diagnosis between 2005 - 2019
* age ≥80 at diagnosis

Exclusion Criteria:

- diagnosis revision at a later timepoint

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with DLBCL
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) death or progression/relapse, progression/relapse or treatment discontinuation. | through study completion, an average of 2 years
  time from diagnosis to death
Progression-free survival (PFS) | through study completion, an average of 2 years
  time from diagnosis to death or progression/relapse
Event-free survival (EFS) | through study completion, an average of 2 years
  defined as time from diagnosis to death or progression/relapse or treatment discontinuation.

SECONDARY OUTCOMES:
Relative Dose intensity | within the treatment period, up to 36 weeks
  Percentage of the dose intensity achieved divided by the intended dose intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University Medical Center, Homburg, Saarland, Germany